CLINICAL TRIAL: NCT06753539
Title: Evaluation of the "Grasp Site" After Peeling of Epiretinal Membranes With Different ILM Forceps - a Prospective Randomized Study
Brief Title: Evaluation of the "Grasp Site" After Peeling of Epiretinal Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Prof. Dr. Oliver Findl, MBA, Sponsor of the study, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIF
Record Dates: First submitted 2024-12-21; First posted 2024-12-31 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Intervention Model Description: Patients were operated on using either an ILM forceps with a laser-modified microstructure on the branches (group A) or a conventional ILM forceps (group B). Patients are randomized to both groups.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ILM sharkskin forceps (Experimental): Patients were operated on using an ILM forceps with a laser-modified microstructure on the branches.
  Interventions: Device: ILM forceps - membrane grasping
- conventional ILM forceps (Active Comparator): Patients were operated on using a conventional ILM forceps with plain surfaces on the branches.
  Interventions: Device: ILM forceps - membrane grasping

INTERVENTIONS:
Device: ILM forceps - membrane grasping — grasping the epiretinal membrane at the starting location, using pinch peeling, is performed with an ILM forceps.

SUMMARY:
The goal of this study is to compare the novel ILM sharkskin forceps with a conventional ILM forceps utilizing iOCT assistance during surgery at this "grasp site". The main questions it aims to answer are:

1. are there differences in grasp attempts between both forceps
2. are there differences in Instrument tissue interactions between both forceps
3. are there differences in postsurgical anatomical and functional outcomes at the grasp site between both forceps.

DETAILED DESCRIPTION:
Epiretinal membranes are a disease of the retinal surface, that may affect visual acuity acuity and cause metamorphopsia, occurring in approximately 20% of the population older than 60 years. Using vitrectomy with membrane peeling, postoperative improvement of visual acuity and metamorphopsia may be achieved in a majority of patients. The surgical method has been used for some time, the first report on the surgical method of vitrectomy with membrane peeling dates back to 1978, and since the introduction of intraoperative optical coherence tomography (iOCT), intraoperative iatrogenically induced changes in retinal tissue can be detected and correlated with postoperative changes. Our group has been able to record "stretching" of the retinal tissue using this technique and has also been able to record the rarely occurring subfoveal and extrafoveal elevations of the ellipsoidal zone due to membrane peeling. These changes did not significantly affect postoperative visual acuity in our study population but did affect the development of postoperative microscotomas. Besides "retinal stretching" during surgery, ILM peeling is shown to be another factor with association of new postoperative microscotomas. New postoperative microscotomas developed in some patients without "retinal stretching" and ILM peeling. Apart from these already known iatrogenic changes, the analysis of the "grasp site" at the "starting point" of epiretinal membrane peeling is of great interest, because at this location, grasping of the epiretinal membrane may be difficult especially in case of an adherent ERM and superficial retinal lesions may be induced.

Diaz et al. demonstrated that there are postoperative changes in the "nerve fiber layer" after ILM peeling, but in that study, no recording of instrument/tissue interactions was performed using iOCT.

The aim of this study is to compare the novel ILM sharkskin forceps with a conventional ILM forceps utilizing iOCT assistance during surgery at this "grasp site".

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic ERM
* Sheduled surgery (vitrectomy with membrane peeling), as defined by vision loss and/or metamorphopsia
* Age 18 and older
* Written informed consent for participation in the study

Exclusion Criteria:

* Macular edema due to other reasons than iERM
* Pregnancy (pregnancy test will be performed in women of reproductive age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
grasp attempts | during surgery
  number of attemps needed for opening the epiretinal membrane during grasping

SECONDARY OUTCOMES:
metamorphopsia | before and 3 months after surgery
  Presence of metamorphopsia is tested with the Amsler grid and M-charts
microscotomata | before and 3 months after surgery
  New deep microscotomata is tested with microperimetry
Thinning of the ganglion cell layer | before and 3 months after surgery
  Thinning of the ganglion cell layer is assessed with optical coherence tomography
Central subfield thickness | before and 3 months after surgery
  Central subfield thickness of the macula is assessed with optical coherence tomography
Best corrected distant visual acuity | before and 3 months after surgery
  Best corrected distant visual acuity is assessed by EDTRS-charts
OCT biomarkers | before surgery
  OCT biomarkers are assessed by optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Leisser, MD, Principal Investigator — Mein Hanusch-Krankenhaus
Locations (1):
- Hanusch Hospital, Department of Ophthalmology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell P, Smith W, Chey T, Wang JJ, Chang A. Prevalence and associations of epiretinal membranes. The Blue Mountains Eye Study, Australia. Ophthalmology. 1997 Jun;104(6):1033-40. doi: 10.1016/s0161-6420(97)30190-0. PMID 9186446
- [Background] Machemer R. [The surgical removal of epiretinal macular membranes (macular puckers) (author's transl)]. Klin Monbl Augenheilkd. 1978 Jul;173(1):36-42. German. PMID 692034
- [Background] Leisser C, Palkovits S, Hienert J, Ullrich M, Zwickl H, Georgiev S, Findl O. Effect of Iatrogenic Traction during Macular Peeling Surgery on Postoperative Microperimetry. Ophthalmic Res. 2021;64(2):273-279. doi: 10.1159/000507633. Epub 2020 Apr 1. PMID 32235121
- [Background] Leisser C, Hackl C, Hirnschall N, Findl O. Effect of Subfoveal and Extrafoveal Hyporeflective Zones due to Iatrogenic Traction during Membrane Peeling for Epiretinal Membranes on Postoperative Outcomes. Ophthalmologica. 2020;243(4):297-302. doi: 10.1159/000505214. Epub 2019 Dec 5. PMID 31801147
- [Background] Diaz RI, Randolph JC, Sigler EJ, Calzada JI. Intraoperative grasp site correlation with morphologic changes in retinal nerve fiber layer after internal limiting membrane peeling. Ophthalmic Surg Lasers Imaging Retina. 2014 Jan-Feb;45(1):45-9. doi: 10.3928/23258160-20131220-06. PMID 24392911